CLINICAL TRIAL: NCT03055442
Title: Altered Myo-inositol/D-chiro-inositol Ratio in Follicular Fluid of Women Undergoing in Vitro Fertilization Has Detrimental Effects on Oocyte and Embryo Quality
Brief Title: Myo-inositol/D-chiro-inositol Ratio in Follicular Fluid
Status: Completed | Type: Observational
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Other Study IDs: MI/DCI_FF
Record Dates: First submitted 2017-02-08; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Women Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Follicular Fluids: Follicular fluids obtained by 8 oocyte donors
  Interventions: Other: Dosage of myo-inositol; Other: Dosage of D-chiro-inositol

INTERVENTIONS:
Other: Dosage of myo-inositol — Quantitative analysis of myo-inositol was performed by gas chromatography-mass spectrometry (GC-MS)
Other: Dosage of D-chiro-inositol — Quantitative analysis of D-chiro-inositol was performed by gas chromatography-mass spectrometry (GC-MS)

SUMMARY:
Considering the importance assumed by follicular microenvironment for a proper oocyte development, this study is a prospective observational clinical trial which aims to evaluate whether the embryo blastocyst quality may be affected by different Myo-inositol (MI) and D-chiro-inositol (DCI) levels in the follicular fluid (FF) of the aspired oocytes. The study includes egg donors and egg receiving couples participating in the oocyte donation program. MI/DCI is calculated in FF and related with blastocyst grade.

ELIGIBILITY:
Inclusion Criteria:

* clear follicular aspirate obtained during oocyte retrieval;
* each specimen of follicular fluid containing only one oocyte.

Exclusion Criteria:

* hyperglycaemic women;
* PCOS women also if euglycaemic;
* diabetic subjects having low concentrations of detectable MI in association with an anomalous MI transport.

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study included 8 egg donors participating in the donation program of IAKENTRO not for the first time, and 11 recipient couples undergoing in vitro fertilization (ICSI).
  Follicular fluid (FF) specimens were analysed.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Myo-inositol concentration (µmol/l) in follicular fluid | 5th day from pick up
  After transvaginal aspiration of oocyte and follicular fluid and subsequent ICSI, at the day 5 the cultured embryos were graded according to Gardner's grading system for blastocysts. Then follicular fluids specimens were divided following the different scores given to the respective blastocysts, and their content in myo-inositol was quantified.
  In each sample of follicular fluid myo-inositol levels were assessed. The quantitative analysis was performed by means of gas chromatography-mass spectrometry (GC-MS) and the values were expressed as µmol/l. This value was related to the respective blastocyst grade.
D-chiro-inositol concentration (µmol/l) in follicular fluid | 5th day from pick up
  After transvaginal aspiration of oocyte and follicular fluid and subsequent ICSI, at the day 5 the cultured embryos were graded according to Gardner's grading system for blastocysts. Then follicular fluids specimens were divided following the different scores given to the respective blastocysts, and their content in D-chiro-inositol was quantified.
  In each sample of follicular fluid D-chiro-inositol levels were assessed. The quantitative analysis was performed by means of gas chromatography-mass spectrometry (GC-MS) and the values were expressed as µmol/l. This value was related to the respective blastocyst grade.

CONTACTS AND LOCATIONS:
Locations (1):
- Iakentro Advanced Medical Centre, IVF Unit, Thessaloniki, Greece

REFERENCES:
- [Background] Chiu TT, Rogers MS, Law EL, Briton-Jones CM, Cheung LP, Haines CJ. Follicular fluid and serum concentrations of myo-inositol in patients undergoing IVF: relationship with oocyte quality. Hum Reprod. 2002 Jun;17(6):1591-6. doi: 10.1093/humrep/17.6.1591. PMID 12042283
- [Background] Carlomagno G, Unfer V, Roseff S. The D-chiro-inositol paradox in the ovary. Fertil Steril. 2011 Jun 30;95(8):2515-6. doi: 10.1016/j.fertnstert.2011.05.027. Epub 2011 Jun 8. PMID 21641593
- [Background] Gardner DK, Lane M, Stevens J, Schlenker T, Schoolcraft WB. Blastocyst score affects implantation and pregnancy outcome: towards a single blastocyst transfer. Fertil Steril. 2000 Jun;73(6):1155-8. doi: 10.1016/s0015-0282(00)00518-5. PMID 10856474
- [Derived] Ravanos K, Monastra G, Pavlidou T, Goudakou M, Prapas N. Can high levels of D-chiro-inositol in follicular fluid exert detrimental effects on blastocyst quality? Eur Rev Med Pharmacol Sci. 2017 Dec;21(23):5491-5498. doi: 10.26355/eurrev_201712_13940. PMID 29243796